CLINICAL TRIAL: NCT06816940
Title: Analysis of Dry Needling Combined With an Exercise Program in the Treatment of Osteoarthritis Knee: Randomized Clinical Trial
Brief Title: Dry Needling and Exercise Program in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Albornoz Cabello (Other)
Responsible Party: Sponsor-Investigator, Manuel Albornoz Cabello, Clinical Professor, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0808-N-22
Record Dates: First submitted 2025-01-14; First posted 2025-02-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Musculoskeletal; Physical Medicine/Rehabilitation; Physiotherapy; Dry needling; Therapeutic exercise
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups, randomly selected (experimental group and control group), of 30 subjects each. Allocation was concealed and it was done by central randomisation by computer (EPIDARcomputer program).The main objective of the study is to observe the resulting data on pain, function, strength and range of motion, in subjects with knee OA, after being treated with a specific exercise program and dry needling technique in the popliteal muscle. All participants will be assessed before carrying out any intervention and after it has been carried out. This assessment will consist of measuring pain, strength, range of motion, and functionality. As for the intervention, both will be treated with a specific exercise program specific for knee osteoarthritis, and only one group will be additionally operated on by the dry needling technique of the popliteal muscle, following the safety criteria of the same.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (Active Comparator): You will be provided exclusively therapeutic exercises protocol to develop in the home setting that you must perform following a daily activity for three weeks.
  Interventions: Other: CONTROL GROUP:
- EXPERIMENTAL GROUP (Experimental): EXPERIMENTAL GROUP: will be provided therapeutic exercises protocol to develop in the home setting that you must perform following a daily activity for three weeks, and rurgery was also performed using the dry needling technique of the popliteal muscle, following its safety criteria.
  Interventions: Other: EXPERIMENTAL GROUP

INTERVENTIONS:
Other: CONTROL GROUP: — will be provided exclusively therapeutic exercises protocol to develop in the home setting that you must perform following a daily activity for three weeks. They will be evaluated before any intervention is carried out
  Arms: CONTROL GROUP
Other: EXPERIMENTAL GROUP — will be provided therapeutic exercises protocol to develop in the home setting that you must perform following a daily activity for three weeks, and rurgery was also performed using the dry needlig
  Arms: EXPERIMENTAL GROUP

SUMMARY:
Osteoarthrosis (OA) is a chronic degenerative disease that affects the joints, knee OA is the most prevalent type, affecting 265 million people worldwide, more than 40% of adults over 45 years of age, being one of the greatest causes of disability, which leads to a decrease in the quality of life of those who suffer from it, and increased medical care and costs.

Currently, clinical guidelines recommend physical exercise as the first line of treatment for knee OA.

Reviews conducted in 2020 observe a low level of evidence regarding dry needling in subjects with OA, suggesting the need for future publications focused on this research problem.

Popliteal muscle involvement is often underestimated in knee pain, however, some authors also suggest that the presence of trigger points in this muscle may represent a cause of diffuse knee pain. Active trigger points in the popliteus have been observed in 17% of people with symptomatic knee OA.

This study aims to evaluate data resulting from pain, function, strength and range of motion, in subjects with OA, after being treated with a specific exercise program and dry needling technique in the popliteal muscle. The subjects will be recruited at a health centre in the city of Seville, and at the Physiotherapy department of the University of Seville.

As this is research with people, the researcherse wanted to be especially attentive to the following ethical aspects: all participants will be informed of the objective of the project and will be asked for written informed consent, their wish not to participate or abandon the project will be respected and they will be guaranteed that the information obtained will be completely anonymous and for use exclusively for the purposes of the research. The informed consent to be given is based on the ethical principles set out in the World Medical Association's 1964 Declaration of Helsinki for medical research involving human subjects. Compliance with the rules of the General Health Law of 1986 and the Basic Law 41/2002 Regulating Patient Autonomy.

1. General Objective To evaluate and compare the resulting data on pain, function, strength, and range of motion in subjects with knee OA after being treated with a specific exercise program; and treated with the same exercise program combined with dry needling technique in the popliteal muscle.

DETAILED DESCRIPTION:
This study will constitute a comparative Randomized Clinical Study (RCT) of two groups with different treatments in subjects diagnosed with knee OA. The control group (CG) will be treated with a specific exercise protocol for knee OA, while the experimental group (EG) will be operated on with the dry needling technique in the popliteal muscle, in addition to performing the same exercise protocol as the CG.

The development of the study will take place over a period of 6 months, starting in March 2024.

A study conducted on cadavers in 2021, shows a safe and effective way to carry out the dry needling technique of the popliteal muscle. With the knee bent at approximately 90°, the needle is inserted from medial to lateral direction into the upper third of the tibia closest to the knee and at an anterior angle toward the posterior aspect of the tibia, remaining as close as possible to the posterior aspect of the tibia bone to a depth that was clinically considered more likely in the popliteal muscle, thus being isolated from the vasculonervous bundle.

Population to be studied The study is designed to be conducted on people of legal age. The target population will be patients diagnosed with knee OA uni or bilaterally, while the eligible population will be all those patients diagnosed with knee OA who attend the Physiotherapy of the "El Cachorro" Health Center in Seville and who can and wish to be part of the study and who meet the inclusion and exclusion criteria.

Subjects diagnosed with uni or bilateral knee OA will be included. Those who do not give their consent to participate, minors and those subjects with knee prostheses, surgical intervention in the area, or treatment in less than 6 months in the study area will be excluded.

Initially, a meeting will be held (in the aforementioned centres) with the patients under study, where they will be informed and any doubts that may arise in relation to the research will be resolved. In addition, the correct adequacy of these to the inclusion and exclusion criteria of our study will be checked. Subsequently, they will be individually given the informed consent prepared expressly for this study, any doubts that may arise regarding it will be resolved and they will be signed. At that time, and individually again, the researchers will proceed to the preparation of the Physiotherapy clinical history where only and exclusively the information necessary for our study will be collected.

The sample will consist of 60 subjects, divided between both groups, diagnosed with knee OA uni or bilaterally, who have given their written consent to participate.

The sample size was obtained for an intergroup interaction with an error α of 95% or less than 0.05, a statistical power Β or 0.95 for two study groups in four measurements with an effect size (F) of 0.20, obtaining a total of 56 participants, 28 in each group, but taking into account a possible loss of 3%. Therefore, the sample will consist of 60 subjects, divided between both groups, diagnosed with knee OA uni or bilaterally, who have given their consent.

The professionals who will perform the intervention of both therapeutic exercise and dry needling are Physiotherapists with more than 10 years of clinical experience and trained in these disciplines.

The variables to be studied will be the same for both groups:

* WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index questionnaire).
* Degree of pain, using the visual analogue scale (VAS).
* DN4 Questionnaire (Douleur Neurophathique 4); Annex V
* Functional disability with the Kujala Score test (Escala de dolor anterior de rodilla).
* Lower Extremity Functional Scale (LEFS).
* Knee flexion and extension joint balance.
* Force using the Daniels scale and dynamometer.
* Fear in relation to pain with TSK-11SV questionnaire (Escala TAMPA de Kinesiophobia)

Data Analysis Plan For data analysis, the SPSS statistical program will be used to obtain the mean, median, maximum, minimum and standard deviation data. The researchers will carry out an analysis of all the variables collected by the scales and the relationships that the different variables have based on Pearson's correlations.

The main objective of the study is to observe the resulting data on pain, function, strength and range of motion, in subjects with knee osteoarthritis, after being treated with a specific exercise program and dry needling technique in the popliteal muscle.

To carry it out, the participants will be divided into two groups, chosen randomly. All participants will be assessed before carrying out any intervention and after it has been carried out. This assessment will consist of measuring pain, strength, range of motion, and functionality.

As for the intervention, both will be treated with a specific exercise program specific for knee osteoarthritis, and only one group will be additionally operated on by the dry needling technique of the popliteal muscle, following the safety criteria of the same.

ELIGIBILITY:
Inclusion Criteria: Subjects diagnosed with uni or bilateral knee OA will be included -

Exclusion Criteria: people who do not give their consent to participate, minors and those subjects with knee replacements, surgical intervention in the area, or treatment in less than 6 months in the study area.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Questionnaire) | Time point 1: They will be assessed before any intervention is carried out
  It is a self-rated questionnaire specifically for patients with osteoarthritis of the hip and knee, which is made up of 24 items divided into 3 scales; pain (5 items), function (17 items), and stiffness (2 items). The answers are coded, being 0 "no difficulty" and 4 "extreme difficulty" to perform the activity (intermediate answers are 1: mild, 2: moderate, 3: severe). The final score is determined by adding the points for pain and function separately, and standardizing them over a range of values from 0 to 100, where 0 represents the best possible state of health and 100 the worst.
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Questionnaire) | Time point 2: It is assessed when the intervention is completed (3 and 6 months after the last session)..
  It is a self-rated questionnaire specifically for patients with osteoarthritis of the hip and knee, which is made up of 24 items divided into 3 scales; pain (5 items), function (17 items), and stiffness (2 items). The answers are coded, being 0 "no difficulty" and 4 "extreme difficulty" to perform the activity (intermediate answers are 1: mild, 2: moderate, 3: severe). The final score is determined by adding the points for pain and function separately, and standardizing them over a range of values from 0 to 100, where 0 represents the best possible state of health and 100 the worst.
EVA (VISUAL ANALOGUE SCALE) | Time point 1:They will be assessed before any intervention is carried out
  A scale used to measure pain that is very similar to a numerical scale. The EVA consists of a 10 cm line with one end with the 0 meaning "no pain" and another end with the 10 indicating "the worst pain imaginable". The patient makes a mark on the line indicating the point that best describes the intensity of their pain. It establishes:
  * Mild pain if the score is less than 3.
  * Moderate pain if it is between 4 and 7.
  * Severe pain if the rating is greater than or equal to 8.
EVA (VISUAL ANALOGUE SCALE) | Time point 2: In GE the subjects will be messured Pre and Post PS Intervention. Both groups is assessed when the intervention is completed (3 and 6 months after the last session)
  A scale used to measure pain that is very similar to a numerical scale. The EVA consists of a 10 cm line with one end with the 0 meaning "no pain" and another end with the 10 indicating "the worst pain imaginable". The patient makes a mark on the line indicating the point that best describes the intensity of their pain. It establishes:
  * Mild pain if the score is less than 3.
  * Moderate pain if it is between 4 and 7.
  * Severe pain if the rating is greater than or equal to 8.
Douleur Neurophatique 4 (DN4) | Time point 1: They will be assessed before any intervention is carried out
  It is a questionnaire consisting of 4 questions with a total of 10 items, which tries to describe symptoms and signs of pain that are evaluated with 1 (yes) or 0 (no) to identify patients who may have neuropathic pain. The lowest total value is 0 and means there is no neuropathic pain. The highest value is 10 for those people who have all the characteristics of neuropathic pain.
  A cut-off point of 4 is set.
Douleur Neurophatique 4 (DN4) | Time point 2: In GE the subjects will be messured Pre and Post PS Intervention. Both groups is assessed when the intervention is completed (3 and 6 months after the last session).
  It is a questionnaire consisting of 4 questions with a total of 10 items, which tries to describe symptoms and signs of pain that are evaluated with 1 (yes) or 0 (no) to identify patients who may have neuropathic pain. The lowest total value is 0 and means there is no neuropathic pain. The highest value is 10 for those people who have all the characteristics of neuropathic pain.
  A cut-off point of 4 is set.
Anterior Knee Pain Scale (KUJALA SCORE) | Time point 1: They will be assessed before any intervention is carried out
  The functional disability, quantified by means of the test: Kujala Score. The 13 items on the scale are used to assess subjective symptoms and functional restrictions. A score can have a minimum of 0 points or a maximum of 100 points. Subjects would receive a score of 100 if they showed no signs of previous knee pain.
Anterior Knee Pain Scale (KUJALA SCORE) | Time point 2: It is assessed when the intervention is completed (3 and 6 months after the last session)
  The functional disability, quantified by means of the test: Kujala Score. The 13 items on the scale are used to assess subjective symptoms and functional restrictions. A score can have a minimum of 0 points or a maximum of 100 points. Subjects would receive a score of 100 if they showed no signs of previous knee pain.
LEFS (Lower Extremity Functional Scale) | Time point 1: They will be assessed before any intervention is carried out
  It is a self-administered 20-item questionnaire that serves to assess the functional capacity of the lower limb. It is a 5-point Likert scale ranging from 0 (extreme difficulty) to 4 (no difficulty). From the scale, a total score is obtained that shows the functionality of the subject's lower limbs. It has a minimum value of 0 points, which indicates that the subject does not have any problems in the functionality of the lower limbs, and a maximum value of 80 points, which indicates severe problems in the functionality of the lower limbs.
LEFS (Lower Extremity Functional Scale) | Time point 2: It is assessed when the intervention is completed (3 and 6 months after the last session)
  It is a self-administered 20-item questionnaire that serves to assess the functional capacity of the lower limb. It is a 5-point Likert scale ranging from 0 (extreme difficulty) to 4 (no difficulty). From the scale, a total score is obtained that shows the functionality of the subject's lower limbs. It has a minimum value of 0 points, which indicates that the subject does not have any problems in the functionality of the lower limbs, and a maximum value of 80 points, which indicates severe problems in the functionality of the lower limbs.
Active and Pasive Knee's Range of Movement | Time point 1: They will be assessed before any intervention is carried out
  In addition an anthropometric study of knee joint range of movement will be performed. Evaluating the Active and Pasive Knee's Range of Movement using universal goniometer measurement. we pay special attention to the possible restrictions in the normal range of motion
Active and Pasive Knee's Range of Movement | Time point 2: In GE the subjects will be messured Pre and Post PS Intervention. Both groups is assessed when the intervention is completed (3 and 6 months after the last session)
  In addition an anthropometric study of knee joint range of movement will be performed. Evaluating the Active and Pasive Knee's Range of Movement using universal goniometer measurement. we pay special attention to the possible restrictions in the normal range of motion
DANIELS SCALE | Time point 1: They will be assessed before any intervention is carried out
  The grades in the manual muscle assessment are obtained in the form of a numerical score ranging from zero (0), which represents the absence of activity, to five (5), which represents a normal response to the test, or as normal as it can be assessed in a manual test. Because this test is performed on the applied movements and not on the muscle individually, so the activity of all the muscles in that movement is evaluated. This scale from 0 to 5 is the most commonly accepted. Each numerical score is accompanied by a word that gives it a qualitative score 5 → normal (N) 4→ good (B) 3 → Regular (R) 2→ Bad (M)
  1→ Low activity (E) 0→ Null (No Activity) (0)
DANIELS SCALE | Time point 2: It is assessed when the intervention is completed (3 and 6 months after the last session)
  The grades in the manual muscle assessment are obtained in the form of a numerical score ranging from zero (0), which represents the absence of activity, to five (5), which represents a normal response to the test, or as normal as it can be assessed in a manual test. Because this test is performed on the applied movements and not on the muscle individually, so the activity of all the muscles in that movement is evaluated. This scale from 0 to 5 is the most commonly accepted. Each numerical score is accompanied by a word that gives it a qualitative score 5 → normal (N) 4→ good (B) 3 → Regular (R) 2→ Bad (M)
  1→ Low activity (E) 0→ Null (No Activity) (0)
TAMPA Scale of Kinesiophobia (TSK-11SV) | Time point 1: They will be assessed before any intervention is carried out
  It is an 11-item questionnaire that is used to assess the patient's fear of suffering the injury again due to movement, i.e., it measures kinesiophobia. The TSK-11 is scored on a 4-point Likert scale, with responses ranging from 1 (strongly disagree) to 4 (strongly agree). The lowest possible score, 11, denotes insignificant or no kinesiophobia. The highest possible score, 44, denotes a severe fear of experiencing pain when moving.
TAMPA Scale of Kinesiophobia (TSK-11SV) | Time point 2: In GE the subjects will be messured Pre and Post PS Intervention. Both groups is assessed when the intervention is completed (3 and 6 months after the last session)
  It is an 11-item questionnaire that is used to assess the patient's fear of suffering the injury again due to movement, i.e., it measures kinesiophobia. The TSK-11 is scored on a 4-point Likert scale, with responses ranging from 1 (strongly disagree) to 4 (strongly agree). The lowest possible score, 11, denotes insignificant or no kinesiophobia. The highest possible score, 44, denotes a severe fear of experiencing pain when moving.

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Escobio Prieto, Lebrija, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agost-Gonzalez A, Escobio-Prieto I, de Los Angeles Cardero-Duran M, Yanez-Alvarez AR, Fernandez-Morales C, Albornoz-Cabello M. Effects of dry needling combined with exercise on knee osteoarthritis at 6 month follow up a randomized clinical trial. Sci Rep. 2025 Dec 18;15(1):44117. doi: 10.1038/s41598-025-27821-0. PMID 41413069